CLINICAL TRIAL: NCT03478982
Title: A Double-Blind, Placebo-Controlled, Inpatient, Dose-Ranging Efficacy Study of Staccato Alprazolam (STAP-001) in Subjects With Epilepsy With a Predictable Seizure Pattern
Brief Title: Inpatient, Dose-Ranging Study of Staccato Alprazolam in Epilepsy With Predictable Seizure Pattern
Acronym: StATES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Engage Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENGAGE-E-001
Record Dates: First submitted 2018-03-07; First posted 2018-03-27 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Staccato Alprazolam 1.0 mg (Experimental): single dose for inhalation
  Interventions: Drug: Staccato Alprazolam
- Staccato Alprazolam 2.0 mg (Experimental): single dose for inhalation
  Interventions: Drug: Staccato Alprazolam
- Placebo (Placebo Comparator): single dose for inhalation
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Staccato Alprazolam — single dose for inhalation
  Other Names: STAP-001
  Arms: Staccato Alprazolam 1.0 mg; Staccato Alprazolam 2.0 mg
Drug: Placebos — single dose for inhalation
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blind, randomized, parallel group, dose-ranging study to investigate the efficacy and clinical usability of STAP-001 in adult (18 years of age and older) subjects with epilepsy with a predictable seizure pattern. These subjects have an established diagnosis of focal or generalized epilepsy with a documented history of predictable seizure episodes. This is an in-patient study. The subjects will be admitted to a Clinical Research Unit (CRU) or Epilepsy Monitoring Unit (EMU) for study participation. The duration of the stay in the in-patient unit will be 2-8 days. One seizure event per subject will be treated with study medication. The duration and timing of the seizure event and occurrence of subsequent seizures will be assessed by the Staff Caregiver(s)1 through clinical observation and confirmed with video electroencephalogram (EEG).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide, personally signed, and dated informed consent to participate in the study or will have a legally authorized representative sign the informed consent on his or her behalf before completing any study related procedures.
2. Male or female ≥ 18 years of age.
3. Has an established diagnosis of focal or generalized epilepsy or focal and generalized epilepsy with a documented history of predictable seizure episodes that includes at least one of the following:

   * Generalized seizure episodes starting with a flurry of absence seizures or myoclonic seizures with a minimum duration of 5 minutes
   * Episodes of a prolonged focal seizure with a minimum duration of 3 minutes
   * Episodes of multiple (≥2) seizures within a 2-hour time period
4. Prior to randomization, has experienced ≥4 seizure episodes with predictable pattern during the last 4 weeks (qualification period) and no more than one week without a predictable seizure episode before entry into the in-patient unit.
5. Female participants (if of child-bearing potential and sexually active) and male participants (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method throughout the study and for 1 week following the end of the study. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm with spermicide,intrauterine device (IUD), surgical sterilization, and progestin implant or injection. Prohibited methods include: the rhythm method, withdrawal, condoms alone, or diaphragm alone.
6. Subject is able to comply by the requirements of the protocol, particularly the requirements and specific Institution policies during the in-clinic stay.

Exclusion Criteria:

1. History or diagnosis of non-epileptic seizures (e.g. metabolic or pseudo-seizures).
2. History of status epilepticus in the 6 months prior to Screening
3. Has a progressive neurological disorder such as brain tumor, demyelinating disease, or degenerative central nervous system (CNS) disease that is likely to progress in the next 3 months
4. Use of strong CYP 3A4 inhibitors; including azole antifungal agents (e.g., etoconazole, itraconazole), nefazodone, fluvoxamine, cimetidine, HIV protease inhibitors (e.g., ritonavir)
5. Has severe chronic cardio-respiratory disease
6. History of HIV-positivity.
7. Pregnant or breast-feeding.
8. Clinically significant renal or hepatic insufficiency (hepatic transaminases >2 times the upper limit of normal (ULN) or creatinine ≥ 1.5 x ULN).
9. History of acute narrow angle glaucoma, Parkinson's disease, hydrocephalus, or history of significant head trauma.
10. Subjects who use medications to treat airways disease, such as asthma or COPD or have any acute respiratory signs/symptoms (e.g., wheezing).
11. Use of any investigational drug within 30 days or 5 half-lives of the investigational drug prior to administration of study medication, whichever is longer
12. A history within the past 1 year of drug or alcohol dependence or abuse.
13. Positive urine screen for drugs of abuse at Screening.(positive Cannabis/Cannabinol results are acceptable if there is a documented history of stable use for medical purposes).
14. Known allergy or hypersensitivity to alprazolam.
15. History of glaucoma.
16. Subjects who currently have an active major psychiatric disorder where changes in pharmacotherapy are needed or anticipated during the study.
17. Hypotension (systolic blood pressure ≤90 mm Hg, diastolic blood pressure ≤50 mm Hg), or hypertension (systolic blood pressure ≥140 mm Hg, diastolic blood pressure ≥100 mm Hg) measured while seated at screening or baseline.
18. Significant hepatic, renal, gastroenterologic, cardiovascular (including ischemic heart disease and congestive heart failure), endocrine, neurologic or hematologic disease.
19. Subjects who, in the opinion of the Investigator, should not participate in the study for any reason, including if there is a question about the stability or capability of the subject to comply with the trial requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Isojarvi, MD, PhD, Study Chair — Engage Therapeutics, Inc.
Locations (67):
- United States (63):
  - UAB Hospital, Birmingham, Alabama
  - University of Arizona, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center - Barrow Neurological Institute, Phoenix, Arizona
  - Clinical Trials Inc, Little Rock, Arkansas
  - Rancho Research Institute Inc., Downey, California
  - UCLA, Los Angeles, California
  - Hoag Hospital, Newport Beach, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Havana Research Institute LLC., Pasadena, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - GW Medical Faculty Associates, Washington D.C., District of Columbia
  - NW FL Clinical Research Group LLC, Gulf Breeze, Florida
  - University of Florida Health Science Center Jacksonville, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Clinical Translational Research Site, Miami, Florida
  - Advanced Pharma Cr, LLC, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Research Institute of Orlando, LLC, Orlando, Florida
  - NeuroMedical Research Institute, Panama City, Florida
  - Center for Rare Neurological Diseases, Norcross, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Health System, New Orleans, Louisiana
  - Maine Medical Center, Scarborough, Maine
  - Mid-Atlantic Epilepsy And Sleep Center, LLC, Bethesda, Maryland
  - Harvard Medical School - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - SRI International, West Bloomfield, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Impact Clinical Trials Las Vegas, Las Vegas, Nevada
  - JFK Medical Center, Edison, New Jersey
  - Institute of Neurology & Neurosurgery at St. Barnabas, Livingston, New Jersey
  - Rutgers University, New Brunswick, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - SUNY Downstate Medical Center - Comprehensive Epilepsy Center, Brooklyn, New York
  - Kaleida Health Oishei Children's Hospital, Buffalo, New York
  - NYU Comprehensive Epilepsy Center, New York, New York
  - Mount Sinai Health System, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Carolinas Neurosciences Institute, Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC, Concord, North Carolina
  - The Promedica-University of Toledo Neuroscience Center, Toledo, Ohio
  - Oregon Health & Science University - Brain Institute - Comprehensive Epilepsy Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Template University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center - Neurology Clinic, Dallas, Texas
  - UT Houston, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Centra Medical Group Neurology Center, Lynchburg, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Multi-Care Institute for Research and Innovation, Tacoma, Washington
- Australia (3):
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred, Melbourne, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
- The Tower, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Derived] French J, Biton V, Dave H, Detyniecki K, Gelfand MA, Gong H, Liow K, O'Brien TJ, Sadek A, DiVentura B, Reich B, Isojarvi J. A randomized phase 2b efficacy study in patients with seizure episodes with a predictable pattern using Staccato(R) alprazolam for rapid seizure termination. Epilepsia. 2023 Feb;64(2):374-385. doi: 10.1111/epi.17441. Epub 2022 Dec 7. PMID 36268811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in March 2018 and concluded in January 2020.
Pre-assignment Details: Participant Flow refers to Enrolled Population.
Groups:
- Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg); Double-blind: Staccato Alprazolam 1.0 mg: Participants received a single dose of alprazolam 1.0 mg as an oral inhalation using the Staccato delivery system at the onset of their predictable seizure episode from Day 1 through the end of Day 7.
- Double-blind: Placebo: Participants received a single dose of placebo matching to alprazolam as an oral inhalation using the Staccato delivery system at the onset of their predictable seizure episode from Day 1 through the end of Day 7.
- Double-blind: Staccato Alprazolam 2.0 mg: Participants received a single dose of alprazolam 2.0 mg as an oral inhalation using the Staccato delivery system at the onset of their predictable seizure episode from Day 1 through the end of Day 7.
Period: Overall Study
Arm/Group | Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg) | Double-blind: Placebo | Double-blind: Staccato Alprazolam 1.0 mg | Double-blind: Staccato Alprazolam 2.0 mg
Started | 11 | 50 | 47 | 48
Enrolled Participants But Not Treated | 3 | 10 | 9 | 10
Intent-to-treat (ITT) Population | 8 | 40 | 38 | 38
Completed | 11 | 50 | 47 | 48
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to Intent-to-treat (ITT) population. ITT population included all participants who had a seizure event and received study drug during the Treatment Period.
Arm/Group | Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg) | Double-blind: Placebo | Double-blind: Staccato Alprazolam 1.0 mg | Double-blind: Staccato Alprazolam 2.0 mg | Total Title
Number analyzed (Participants) | 8 | 40 | 38 | 38 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (14.51) | 33.1 (9.80) | 34.8 (11.18) | 33.5 (11.74) | 34.7 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 20 | 21 | 26 | 75
  Male | 0 | 20 | 17 | 12 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 1 | 3
  Black or African American | 0 | 8 | 2 | 2 | 12
  Native Hawaiian / Pacific Islander | 2 | 2 | 0 | 1 | 5
  White | 4 | 26 | 36 | 28 | 94
  Declined to Answer | 0 | 1 | 0 | 2 | 3
  Other | 2 | 0 | 0 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Each Treatment Group Achieving Seizure Activity Cessation Within 2 Minutes and no Recurrent Seizure Within 2 Hours
Description: Percentage of participants with onset of a predictable seizure through 2 minutes post dosing with study drug and no recurrence of seizure activity within 2 hours were reported for each treatment group based on clinical observation.
Time Frame: 2 hours post-dosing on dosing day
Population: The Modified Intent-to-treat (mITT) population consisted of all participants who had a seizure event, received study drug, and had at least one evaluation after study drug administration.
Measure: Number; unit: percentage of participants
Arm/Group | Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg) | Double-blind: Placebo | Double-blind: Staccato Alprazolam 1.0 mg | Double-blind: Staccato Alprazolam 2.0 mg
Number analyzed (Participants) | 8 | 40 | 38 | 38
percentage of participants | 62.5 | 42.5 | 65.8 | 65.8
Statistical Analysis 1: Comparison: Double-blind: Placebo vs Double-blind: Staccato Alprazolam 1.0 mg; Test type: Superiority; p = 0.0392, Chi-squared; Difference in percentage = 23.3, 95% CI 2-sided [1.8 to 44.8]
Statistical Analysis 2: Comparison: Double-blind: Placebo vs Double-blind: Staccato Alprazolam 2.0 mg; Test type: Superiority; p = 0.0392, Chi-squared; Difference in percentage = 23.3, 95% CI 2-sided [1.8 to 44.8]

2. Secondary Outcome: Percentage of Participants With Seizure Episode Severity Assessed by Seizure Episode Severity Scale
Description: Severity of on study seizure episode compared to previously experienced seizures was assessed with Seizure Episode Severity Scale. It is a 5-point scale with range from 1 to 5, where 1 indicates much worse than and 5 indicates much better than.
Time Frame: 6 hours post-dosing on dosing day
Population: The mITT population consisted of all participants who had a seizure event, received study drug, and had at least one evaluation after study drug administration.
Measure: Number; unit: percentage of participants
Arm/Group | Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg) | Double-blind: Placebo | Double-blind: Staccato Alprazolam 1.0 mg | Double-blind: Staccato Alprazolam 2.0 mg
Number analyzed (Participants) | 8 | 40 | 38 | 38
percentage of participants
  Much worse than | 0 | 2.5 | 0 | 0
  Worse than | 0 | 5.0 | 2.6 | 5.3
  Same as | 12.5 | 42.5 | 57.9 | 55.3
  Better than | 50.0 | 35.0 | 18.4 | 28.9
  Much better than | 25.0 | 7.5 | 15.8 | 5.3
  Not done | 12.5 | 7.5 | 5.3 | 5.3

3. Secondary Outcome: Percentage of Participants With Use of Rescue Medication
Description: Percentage of participants with use of rescue medication to stop a seizure episode at the discretion of the principal investigator were reported.
Time Frame: 2 hours post-dosing on dosing day
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg) | Double-blind: Placebo | Double-blind: Staccato Alprazolam 1.0 mg | Double-blind: Staccato Alprazolam 2.0 mg
Number analyzed (Participants) | 8 | 40 | 38 | 38
percentage of participants | 0 | 7.5 | 15.8 | 7.9

4. Secondary Outcome: Percentage of Participants With Secondary Generalization (Evolution to a Complex Partial Seizure and/or a Generalized Tonic-Clonic Seizure)
Description: Percentage of participants who had seizures that evolved to a complex partial seizure and/or a generalized tonic-clonic seizure were reported.
Time Frame: 24 hours post-dosing on dosing day
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg) | Double-blind: Placebo | Double-blind: Staccato Alprazolam 1.0 mg | Double-blind: Staccato Alprazolam 2.0 mg
Number analyzed (Participants) | 8 | 40 | 38 | 38
percentage of participants | 12.5 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From Screening up to 12 weeks
Description: The Safety Population included all participants who received study drug during the Treatment Period from either Open-label Feasibility or Double-blind Phase.
Arm/Group | Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg) | Double-blind: Placebo | Double-blind: Staccato Alprazolam 1.0 mg | Double-blind: Staccato Alprazolam 2.0 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/40 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/40 | 1/38 | 0/38
Other Adverse Events (participants affected / at risk) | 3/8 | 10/40 | 14/38 | 19/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg) (N=8) | Double-blind: Placebo (N=40) | Double-blind: Staccato Alprazolam 1.0 mg (N=38) | Double-blind: Staccato Alprazolam 2.0 mg (N=38)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure cluster (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label: Staccato Alprazolam (STAP-001) 1.0 Milligram (mg) (N=8) | Double-blind: Placebo (N=40) | Double-blind: Staccato Alprazolam 1.0 mg (N=38) | Double-blind: Staccato Alprazolam 2.0 mg (N=38)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 7 (8) | 4 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 6 (6) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (3)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 7 (7)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine phosphorus (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03478982/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03478982/SAP_001.pdf